CLINICAL TRIAL: NCT01650948
Title: Evaluation of Genetic Variants in Patients Under Treatment for Choroidal Neovascular (CNV) Age-related Macular Degeneration (AMD), Receiving Intravitreal antiVEGF Injections to Evaluate the Association Between Genetic Load and Phenotypes Associated With More Aggressive Forms of Disease.
Brief Title: Genetic Load and Phenotype in Aggressive AMD
Acronym: RPED Genetics
Status: Completed | Type: Observational
Sponsor: Sequenom, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SQNM-AMD-106
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Age-related Macular Degeneration
Keywords: age-related macular degeneration; AMD
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA samples and remnants will be destroyed after analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- AMD subjects with GA and/or RPED: All subjects will have AMD and GA and/or RPED.
  Interventions: Device: RetnaGene AMD LDT
- AMD subjects with CNV alone: All subjects will have the CNV form of AMD only.
  Interventions: Device: RetnaGene AMD LDT

INTERVENTIONS:
Device: RetnaGene AMD LDT

SUMMARY:
Patients with AMD will provide cheek cell samples to determine if their is a correlation between genotype (DNA markers) and phenotype (the type of AMD the patient has).

DETAILED DESCRIPTION:
This study seeks to test individuals who have already progressed to various forms of AMD to evaluate correlations between genetic markers and particular features of AMD including geographic atrophy and pigment epithelial detachments. We hypothesize that patients with more aggressive forms of AMD will have a higher genetic burden contributed by markers in ARMS 2, Complement Factor H (CFH), Complement component 3 (C3), Complement component 2 (C2) , Factor B (FB), or other genetic polymorphisms associated with CNV.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female 50 years of age and older
* Subject provides a signed and dated informed consent
* Subject agrees to provide two buccal swabs in accordance with this protocol
* Diagnosis of CNV secondary to AMD in at least one eye

Exclusion Criteria:

* Previous sample donation under this protocol
* Presence of retinal disease involving the photoreceptors and/or outer retinal layers other than AMD loss such as high myopia, retinal dystrophies, central serous retinopathy, vein occlusion, diabetic retinopathy and uveitis or similar outer retinal diseases which have been present prior to the age of 50.
* Opacities of the ocular media, limitations of pupillary dilation or other problems sufficient to preclude adequate imaging of the posterior segment.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AMD who are or have been treated with anti-VEGF therapy
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The identification of individual genetic markers or a quantitative measure of total genetic burden found to be significantly associated (p value <0.05) with group classification (CNV only versus CNV with GA and/or RPED). | 1 day

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Pacific Eye Associates, San Francisco, California
  - Retina Associates of Kentucky, Lexington, Kentucky
  - Tennessee Retina, Nashville, Tennessee